CLINICAL TRIAL: NCT03472859
Title: Treatment of Dilated Blood Vessels on the Cheeks With a New Yellow Laser and a Traditional Green Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R17111
Record Dates: First submitted 2018-02-26; First posted 2018-03-21 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-02

CONDITIONS: Telangiectasia; Rosacea
Keywords: laser; lasers; KTP; semiconductor; tgs; rosacea; telangiectasia
MeSH Terms: conditions — Telangiectasis; Rosacea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Split-face group 1 (Experimental): In group 1 the left side of the face will be treated with KTP and right side with PHOTOLASE.
  Interventions: Device: PHOTOLASE; Device: KTP
- Split-face group 2 (Experimental): In group 2 the right side of the face will be treated with KTP and left side with PHOTOLASE.
  Interventions: Device: PHOTOLASE; Device: KTP

INTERVENTIONS:
Device: PHOTOLASE — This is the investigational yellow laser (PHOTOLASE)
  Other Names: yellow laser
Device: KTP — This is the traditional green laser (KTP)
  Other Names: green laser

SUMMARY:
The goal is to compare a novel yellow laser, based on semiconductor technology, with traditional green laser, in the treatment of cheek telangiectasias. The trial design is randomized split-face double-blinded study with 20-30 volunteers. The improvement will be assessed using a 7-point Telangiectasia Grading Scale.

DETAILED DESCRIPTION:
Trial design: The study is a comparative randomized split-face double-blinded study without a control group. It enables a comparison between two lasers; namely the KTP laser and the investigational PHOTOLASE laser. The split-face design eliminates the individual biases and the randomization eliminates the possible small variations in the symmetry of the telangiectasias on the face. The double-blinded assessment eliminates the physicians' and the subjects' subjective and objective bias.

Methods: The subjects will be treated with a 532-nm green KTP laser and a 585-nm yellow PHOTOLASE laser; different laser on each side of a face. A total of one or two treatments will be given based on the response of the first treatment. The improvement of subjects' telangiectasia will be graded after the final treatment according to a 7-point Telangiectasia Grading Scale (TGS) by a blinded physician using images taken with Visia imaging system. The usability, reliability and treatment characteristics of PHOTOLASE laser will be qualitatively assessed by the treating physicians (not blinded).

Objectives: The primary objective is to assess how the PHOTOLASE laser compares to the KTP laser in the treatment of facial telangiectasia in terms of the treatment outcomes. The secondary objective is to assess the usability, reliability and treatment characteristics of the PHOTOLASE laser from the perspective of the user.

ELIGIBILITY:
Inclusion Criteria:

* The subjects are required to be Finnish speaking adults with symmetrical facial telangiectasia, volunteering to participate in the clinical trial.
* The subjects have to have a Fitzpatrick skin phototype I-IV.

Exclusion Criteria:

* pregnancy
* lactation
* hemophilic condition
* Fitzpatrick skin phototype V-VI
* drug or alcohol abuse
* subjects who are under guardianship
* subjects with significant tanning less than 6 weeks prior to the treatment day.
* unbalanced basic diseases, such as diabetes, heart disease, cancer etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-06-09 (Actual); Study Completion 2018-06-09 (Actual)

PRIMARY OUTCOMES:
TGS change | Before treatment and 1-2 months after the intervention.
  Telangiectasia grading scale will be used to assess improvement of telangiectasia and erythema. The range of TGS is -1 to 5, where -1 means worsening of the condition, 0 means no change, 1 means 0-25% improvement, 2 means 25-50% improvement, 3 means 50-75% improvement, 4 means 75-100% improvement and 5 means total clearance.

SECONDARY OUTCOMES:
VAS pain measurement | Immediately after intervention.
  Visual Analogue Scale will be used to measure the amount of pain after the intervention. The range is 0.0 - 10.0, where 0 means no pain and 10 means worst imaginable pain. The results will be reported as a mean value and range for yellow laser and green laser separately.
Amount of treatment-related adverse effects using a 4-point scale. | Immediately after treatment and 2-3 days after treatment.
  The amount of erythema, crusting, edema, purpura and blisters will be assessed separately on both sides of the face. The measurement range is 0-3, where 0 means no symptoms, 1 means mild symptoms, 2 means moderate symptoms and 3 means severe symptoms. The results will be reported as a mean value for yellow laser and green laser separately.

CONTACTS AND LOCATIONS:
Overall Officials: Mircea Guina, Prof, Study Director — Tampere University of Technology, ORC
Locations (1):
- Epilaser Oy, Lempäälä, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No